CLINICAL TRIAL: NCT01361997
Title: Comparative Study of 70% Isopropyl Alcohol Against 2% Chlorhexidine- 70% Isopropyl Alcohol as Antiseptics to Prevent Hemoculture's Contamination
Brief Title: Isopropyl Alcohol Against Chlorhexidine - Isopropyl Alcohol as Antiseptics to Prevent Hemoculture's Contamination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Alejandro E. Macias, Full-time professor, Universidad de Guanajuato
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2011HRAEB001
Record Dates: First submitted 2011-05-23; First posted 2011-05-27 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2012-08

CONDITIONS: Infectious Diseases
Keywords: Antiseptics; Hemoculture contamination; Anti-infecting agents, local
MeSH Terms: conditions — Communicable Diseases | interventions — Chlorhexidine; 2-Propanol; Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine in isopropyl alcohol (Experimental): This arm is composed of 545 hospitalized patients with suspected blood stream infection, to test 2% chlorhexidine gluconate in 70% isopropyl alcohol.
  Interventions: Biological: chlorhexidine in isopropyl alcohol
- Isopropyl alcohol (Experimental): This arm is composed of 572 hospitalized patients with suspected blood stream infection, to test 70% isopropyl alcohol.
  Interventions: Biological: Isopropyl alcohol

INTERVENTIONS:
Biological: chlorhexidine in isopropyl alcohol — When a hemoculture is ordered, the laboratory technician will prepare the necessary materials for venipuncture. Previously the technician must take randomly a sealed envelope, where will be writing the antiseptic to be used for antisepsis. The technician will select a site for venipuncture, preferably in the forearm, and will do the antisepsis in the site selected, letting act the substance for 45 seconds. After this procedure, the venipuncture shall be done. The sample will be cultured for 120 hours at 35 +/- 2°C.
  Other Names: Chloraprep, Enturia Inc., Texas.; BacT/ALERT FA, Biomérieux Inc., North Carolina.
  Arms: Chlorhexidine in isopropyl alcohol
Biological: Isopropyl alcohol — When a hemoculture is ordered, the laboratory technician will prepare the necessary materials for venipuncture. Previously the technician must take randomly a sealed envelope, where will be writing the antiseptic to be used for antisepsis. The technician will select a site for venipuncture, preferably in the forearm, and will do the antisepsis in the site selected, letting act the substance for 45 seconds. After this procedure, the venipuncture shall be done. The sample will be cultured for 120 hours at 35 +/- 2°C.
  Other Names: Alcohol Swabs, BD, Madrid.; BacT/ALERT FA, Biomérieux Inc., North Carolina.
  Arms: Isopropyl alcohol

SUMMARY:
The purpose of this study is to determinate if 70% isopropyl alcohol is not inferior preventing contamination of peripheral hemocultures, compared with 2% chlorhexidine in 70% isopropyl alcohol.

DETAILED DESCRIPTION:
The develop of contaminants in blood cultures is a problem of great impact to health institutions and patients, as they represent a waste of resources, and additionally increases the patient's hospital stay. The principal source of contaminant is the bacteria in the skin flora, so the greatest way to improve the sensibility of this test is to do an optimal skin antisepsis. It has been reported that 2% chlorhexidine gluconate in 70% isopropyl alcohol is superior that other skin disinfectants, and that 70% isopropyl alcohol has a high efficacy reducing the presence of bacteria on the skin, so both antiseptics are good options for skin antisepsis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected blood stream infection.
* Patients allocated in admission, hospitalization and intensive care units.

Exclusion Criteria:

* Patients with a single peripheral hemoculture.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1102 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Determine if 70% isopropyl alcohol is not inferior preventing contamination of peripheral hemoculture, compared with 2% chlorhexidine in 70% isopropyl alcohol. | 120 hours
  It will determine the growth of contaminating germs in hemocultures taken with each antiseptic tested.

SECONDARY OUTCOMES:
Determine the rate of contamination of each antiseptic used. | 1 year
  It will determine the rate of contamination at the date of primary completion and the date of study completion. We will consider contaminants the development of Staphylococcus coagulase negative and gram positive bacilli.
Description of the most frequent bacterial contaminants. | 1 year
  It will determine the rate of contamination at the date of primary completion and the date of study completion. We will consider contaminants the development of Staphylococcus coagulase negative and gram positive bacilli.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro E. Macias, M. D., Principal Investigator — Universidad de Guanajuato
Locations (1):
- University of Guanajuato School of Medicine, León, Guanajuato, Mexico